CLINICAL TRIAL: NCT02556099
Title: EXpanding Treatment for Existing Neurological Disease (EXTEND)
Brief Title: EXTEND EXpanding Treatment for Existing Neurological Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Caribbean Institute for Health Research (CAIHR) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2014-2875 EXTEND
Record Dates: First submitted 2015-05-18; First posted 2015-09-22 (Estimated); Last update posted 2025-08-22 (Actual); Status verified 2025-07

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — Hydroxyurea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hydroxyurea Treatment (Experimental): Hydroxyurea will be administered once daily by mouth. Participants will be monitored monthly to maximum tolerated dose and quarterly thereafter with periodic clinical evaluations, laboratory tests, and transcranial doppler examinations every 6 months.
  Interventions: Drug: Hydroxyurea

INTERVENTIONS:
Drug: Hydroxyurea — drug to be administered

SUMMARY:
The primary goal of the Phase II EXTEND trial is to investigate the effects of open-label hydroxyurea treatment, escalated to maximum tolerated dose, for children with Sickle Cell Anemia and either conditional (170 - 199 cm/sec) or abnormal (≥200 cm/sec) Transcranial Doppler velocities. The primary endpoint will be measured after 18 months of hydroxyurea but treatment will continue until a common study termination date.

DETAILED DESCRIPTION:
Hydroxyurea treatment: Participants will be treated with open-label hydroxyurea, available as 500 mg capsules or liquid (100 mg/mL). Hydroxyurea will be administered once daily by mouth. Participants will be monitored monthly to maximum tolerated dose and quarterly thereafter with periodic clinical evaluations, laboratory tests, and transcranial doppler examinations every 6 months.

Hydroxyurea will be titrated to the maximum tolerated dose as defined by mild marrow suppression, even if the participant has clinical well-being at a lower hydroxyurea dose. The target absolute neutrophil count (ANC)on hydroxyurea therapy will be < 3.0 x 109/L, but the marrow suppression should also include reduction of the reticulocyte count. Hydroxyurea dosing will commence at 20 mg/kg/day. Dose escalation will occur in 5 mg/kg/day increments, adjusting every 8 weeks unless dose-limiting hematological toxicity occurs (defined as ANC < 1.0 x 109/L, hemoglobin concentration < 5 gm/dL or 20% below baseline, absolute reticulocyte count < 80 x 109/L unless hemoglobin concentration >9.0 gm/dL, or platelet count < 80 x 109/L) or the target neutropenia (ANC < 3.0 x 109/L) is achieved. Based on pilot data and experience in other clinical trials, most pediatric participants require hydroxyurea doses of 20-30 mg/kg/day to reach this target absolute neutrophil count .

After reaching maximum tolerated dose, minor hydroxyurea dose adjustments can be made periodically, as necessary based on weight changes and blood counts, to maintain the optimal laboratory response and to prevent dose-related toxicity. If the absolute neutrophil count (ANC) rises above the target range on 2 consecutive visits, compliance will be reinforced and the dose may be adjusted by 2.5 mg/kg/day at eight week intervals to a maximum of 35 mg/kg/day or 2000 mg/day. For hydroxyurea dosing, the current body weight will be used, with dose escalations guided by hematological toxicity. Hydroxyurea will be reduced or even temporarily discontinued for hematological toxicities, e.g., ANC < 1.0 x 109/L, hemoglobin < 5.0 gm/dL, or 20% below baseline, absolute reticulocyte count < 80 x 109/L unless hemoglobin concentration > 9.0 gm/dL, or platelets < 80 x 109/L.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric participants with a severe form of sickle cell anemia (HbSS, HbSβ0 thalassemia, HbSD, HbSOArab)
2. Age: ≥ 2 and ≤ 17 years of age, at the time of enrollment
3. Time-averaged maximum velocity (TAMV) TCD Velocity in the conditional (170 - 199 cm/sec) or abnormal (≥200 cm/sec) range by Transcranial Doppler ultrasonography examination within 6 months of enrollment, abnormal or conditional TCD velocity and currently on commercial hydroxyurea for primary stroke prevention, or previously enrolled in SCATE, a previous stroke with abnormal or conditional TCD prior to stroke event.
4. Parent or guardian willing and able to provide informed consent and child gives assent
5. Ability to comply with study related treatments, evaluations, and follow- up visits

Exclusion Criteria:

1. Inability to take or tolerate daily oral hydroxyurea, including

   * Known allergy to hydroxyurea therapy
   * Known positive serology to HIV infection
   * Known malignancy
   * Current lactation
2. Abnormal historical laboratory values (most recent pre-enrollment values unless previously enrolled in SCATE):

   * Hemoglobin concentration < 6.0 gm/dL
   * Absolute reticulocyte count < 100 x 109/L with a hemoglobin concentration < 8.0 gm/dL
   * White Blood Cell (WBC) count < 3.0 x 109/L
   * Absolute neutrophil count (ANC) < 1.0 x 109/L
   * Platelet count < 100 x 109/L
3. Use of therapeutic agents for sickle cell disease (e.g., hydroxyurea, arginine, decitabine, magnesium, chronic transfusions) within 3 months of enrollment unless they have an abnormal TCD velocity and receive commercial hydroxyurea for primary stroke prevention or were previously enrolled in the SCATE study or for secondary stroke prevention in a child with a previous stroke.
4. Current participation in other therapeutic clinical trials, except SCATE
5. Known serum creatinine more than twice the upper limit for age AND

   * 1.0 mg/dL
6. Any condition or chronic illness, which in the opinion of the clinical investigator makes participation ill-advised
7. Pregnancy (for post-menarchal females only)
8. Erythrocyte transfusion within the past 2 months
9. Previous stem cell transplant or other myelosuppressive therapy (unless they have an abnormal TCD velocity and receive commercial hydroxyurea for primary stroke prevention or for secondary stroke prevention in a child with a previous stroke or were previously enrolled in SCATE)

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 43 (Actual)
Dates: Start 2014-08; Primary Completion 2023-01-16 (Actual); Study Completion 2023-01-16 (Actual)

PRIMARY OUTCOMES:
Maximum Time-Averaged Mean velocity (TAMV) on TCD exam | 18 months
  The primary endpoint of the EXTEND trial is the maximum Time-Averaged Mean velocity (TAMV) on TCD exam performed after 18 months of hydroxyurea treatment, compared to pre-treatment velocity.

SECONDARY OUTCOMES:
Serial TCD velocities | Screening, Baseline, month 6, month 12, month 18
  Serial TCD velocities will be measured every 6 months during the trial. The outcome measure will be the highest TAMV obtained in the main intracranial arteries: middle cerebral artery (MCA), internal carotid artery (ICA), or internal carotid bifurcation (Bif). The TCD velocities at 6-month intervals of hydroxyurea treatment, compared to the baseline pre-treatment TCD values, will describe the potential efficacy of hydroxyurea to reduce elevated TCD velocities.
The cumulative incidence of neurological events | Screening/Baseline and approximately 3 years after the first enrollment
  The cumulative incidence of neurological events, which include both stroke and non-stroke neurological events, will be determined over the treatment period. All potential stroke events will be centrally reviewed by an independent MCC-appointed medical monitor.
Cumulative Incidence of Non-Neurological Events | Screening/Baseline and approximately 3 years after the first enrollment
  The cumulative incidence of non-neurological sickle cell-related events, including vaso-occlusion and splenic sequestration, will be estimated over the treatment period.
Quality of Life Assessment | Baseline, 18 months, and approximately 3 years after the first enrollment
  Quality of Life will be measured at baseline, after 18 months of hydroxyurea treatment, and at study exit using the PedsQL 4.0. The outcome measure will be the overall score obtained by this Quality of Life instrument, as scored by the parent or caregiver. This Quality of Life instrument has been previously standardized and validated in children with chronic illness. A sickle cell disease-specific PedsQL instrument may also be used if available.
Neuropsychological Assessment | Baseline, after 18 months
  Neurodevelopment will be measured at baseline and after 18 months of hydroxyurea treatment, using a standardized neuropsychological assessment tool such as the Wechsler assessments of intelligence. The neuropsychological assessment will be administered as developmentally appropriate, and thus may not be administered to all participants. The outcome measure will be the overall score obtained by this tool.

CONTACTS AND LOCATIONS:
Overall Officials: Russell Ware, MD, PhD, Principal Investigator — Cincinnati Children's
Locations (1):
- Sickle Cell Unit, Kingston, Jamaica

REFERENCES:
- [Derived] Power-Hays A, McElhinney KE, Williams TN, Mochamah G, Olupot-Olupot P, Paasi G, Reid ME, Rankine-Mullings AE, Opoka RO, John CC, McGann PT, Quinn CT, Punt NC, Smart LR, Stuber SE, Latham TS, Vinks AA, Ware RE. Hydroxyurea pharmacokinetics in children with sickle cell anemia across different global populations. Blood Adv. 2026 Jan 27;10(2):418-427. doi: 10.1182/bloodadvances.2025017254. PMID 41026975
- [Derived] Rankine-Mullings AE, Little CR, Reid ME, Soares DP, Taylor-Bryan C, Knight-Madden JM, Stuber SE, Badaloo AV, Aldred K, Wisdom-Phipps ME, Latham T, Ware RE. EXpanding Treatment for Existing Neurological Disease (EXTEND): An Open-Label Phase II Clinical Trial of Hydroxyurea Treatment in Sickle Cell Anemia. JMIR Res Protoc. 2016 Sep 12;5(3):e185. doi: 10.2196/resprot.5872. PMID 27619954